CLINICAL TRIAL: NCT02429440
Title: Adjuvant Antigen Specific Immunotherapy in Patients With Advanced Renal Cell Carcinoma Using Tumor Associated Peptides
Acronym: UroRCC
Status: Unknown | Phase: Phase 1 / Phase 2 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: University Hospital Tuebingen (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 231/2004
Record Dates: First submitted 2015-04-14; First posted 2015-04-29 (Estimated); Last update posted 2017-08-17 (Actual); Status verified 2017-08

CONDITIONS: Renal Cell Cancer; Advanced Renal Cell Cancer
MeSH Terms: conditions — Carcinoma, Renal Cell | interventions — Protein Subunit Vaccines; Granulocyte-Macrophage Colony-Stimulating Factor; montanide ISA 51

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Study Arm 1 (Experimental): Intradermal application of peptide vaccine in combination with Granulocyte Macrophage Colony Stimulating Factor (GM-CSF)
  Interventions: Biological: peptide vaccine; Drug: Granulocyte Macrophage Colony Stimulating Factor
- Study Arm 2 (Active Comparator): Intradermal application of peptide vaccine with Montanide ISA-51
  Interventions: Biological: peptide vaccine; Drug: Montanide ISA-51

INTERVENTIONS:
Biological: peptide vaccine — subcutaneous
Drug: Granulocyte Macrophage Colony Stimulating Factor — intradermal
  Other Names: GM-CSF
  Arms: Study Arm 1
Drug: Montanide ISA-51 — subcutaneous
  Arms: Study Arm 2

SUMMARY:
Clinical Phase I/II study to investigate the feasibility and tolerability of synthetic adjuvant peptide immunisation in combination with immune adjuvants (granulocyte macrophage colony stimulating factor; Montanide ISA-51) in patients with advanced renal cell cancer (RCC).

ELIGIBILITY:
Inclusion Criteria:

* Advanced renal cell carcinoma clinical stage T3 or T4, N0, M0
* N+, M0
* M1 (after complete metastasectomy)
* ECOG performance status 0 or 1
* age >18 years
* at least 4 weeks since last administration of radiation- or chemotherapy
* Serum levels of bilirubin <2 mg/dl, creatinine<2mg/dl

Exclusion Criteria:

* detectable distant metastasis in radiological imaging (M1)
* patients unable to consent
* severe cardiopulmonary disorder (NYHA >= 3)
* presence of secondary malignancy
* Immunosuppressive medication (last application of glucocorticoids > 4 weeks)
* seizure
* pregnancy
* simultaneous participation in other active or passive immunisation treatment

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2005-05; Primary Completion 2017-10 (Estimated); Study Completion 2018-06 (Estimated)

PRIMARY OUTCOMES:
Tolerability | Day 0-365
  Tolerability, as measured by number of Participants with Adverse Events

SECONDARY OUTCOMES:
All Cause Mortality | 60 Months
  All cause Mortality, as measured as length of Overall Survival
Progression-free Survival | 36 Months
  Progression-free Survival, as measured as time to radiographic progression
Immune Response | Day 0-365
  Immune Response, as as measured by in vitro and in vivo T cell response on day 0 and day 70. In selected cases additional immune response evaluation might be applicable.

CONTACTS AND LOCATIONS:
Overall Officials: Arnulf Stenzl, Prof., Principal Investigator — University of Tübingen, Department of Urology